CLINICAL TRIAL: NCT06956599
Title: Clinical Investigation of Hypersensitivity Reduction Efficacy: 5% Potassium Nitrate Toothpaste Compared to Colgate Cavity Protection Toothpaste
Brief Title: Hypersensitivity Reduction Efficacy: 5% Potassium Nitrate Toothpaste Compared to Colgate Cavity Protection Toothpaste
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRO-2025-04-SEN-PNT-YPZ
Record Dates: First submitted 2025-04-25; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Dentin Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Toothpaste (Experimental): Subjects will be instructed to brush their teeth with their assigned test dentifrice and toothbrush twice daily
  Interventions: Drug: test toothpaste
- Control toothpaste (Active Comparator): Subjects will be instructed to brush their teeth with their assigned test dentifrice and toothbrush twice daily
  Interventions: Drug: Control toothpaste

INTERVENTIONS:
Drug: test toothpaste — A commercially available fluoride toothpaste
  Arms: Test Toothpaste
Drug: Control toothpaste — A commercially available fluoride toothpaste
  Arms: Control toothpaste

SUMMARY:
Assess the clinical efficacy of 5% Potassium Nitrate Toothpaste (Colgate-Palmolive Company, New York, NY, USA) on providing dentinal hypersensitivity relief (tactile and air blast) in comparison to Colgate Cavity Protection Toothpaste (Colgate-Palmolive Company, New York, NY, USA) over an eight-week period

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, ages 18-70, inclusive.- Availability for the eight-week duration of the study.
* Two sensitive teeth, which must be anterior to the molars, and demonstrate cervical erosion/abrasion or gingival recession.
* Qualifying response to tactile stimuli (Yeaple probe) as defined by a score between 10-50 gms. of force.
* Qualifying response to the air blast stimuli as defined by a score of 2 or 3 on the Schiff Cold Air Sensitivity Scale.
* Subjects need to satisfy the qualifying response to stimuli for both the parameters assessed (tactile or air) on two teeth to be entered into the study.
* Good general health with no known allergies to products being tested.
* Use of a non-desensitizing dentifrice for three months prior to entry into the study.
* Signed Informed Consent Form

Exclusion Criteria:

* Gross oral pathology, chronic disease, or history of allergy to test products.
* Advanced periodontal disease or treatment for periodontal disease (including surgery) within the past twelve months.
* Sensitive teeth with a mobility greater than one.
* Teeth with extensive/defective restorations (including prosthetic crowns), suspected pulpitis, caries, cracked enamel, or used as abutments for removable partial dentures.
* Current use of anticonvulsants, antihistamines, antidepressants, sedatives, tranquilizers, anti-inflammatory drugs, or daily use of analgesics.
* Participation in a desensitizing dentifrice study or regular use of a desensitizing dentifrice within the past three months.
* Current participation in any other clinical study.
* Pregnant or lactating subjects.
* Allergies to oral care products, personal care consumer products, or their ingredients.
* Medical condition which prohibits not eating/drinking for 4 hours.
* Use in the past of the three test dentifrices.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
tactile sensitivity | baseline and 4 weeks, 8 week measurement
  tactile stimulation is measured by the Yeaple Electronic Force Sensing Probe

SECONDARY OUTCOMES:
air blast sensitivity | baseline and 4 weeks, 8 week measurement
  air blast sensitivity is delivered by a standard dental unit syringe at a measured temperature of 19-21°C (70°F [± 3°F]) [sensitivity will be defined by a score of 2 or 3 on the Schiff Cold Air sensitivity scale Air Sensitivity Scale